CLINICAL TRIAL: NCT03124173
Title: Cognitive Control of Language and Frontal Cortex
Brief Title: Cognitive Control of Language
Acronym: LANGUAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0684
Record Dates: First submitted 2017-03-09; First posted 2017-04-21 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: fMRI; cingulate cortex; adaptation; frontal cortex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral Tasks (Other): Each subject will conduct 4 sessions, i.e. a training session and three fMRI sessions. The first session will consist in training the subject to carry out the different behavioral tasks that he will then have to perform during the sessions of fMRI.
  Interventions: Other: Training session; Other: First fMRI session; Other: Second fMRI session; Other: Third session of fMRI

INTERVENTIONS:
Other: Training session — The subjects will be trained to realize several versions of a learning task of conditional visuo-motor associations.
Other: First fMRI session — In this session (involving a condition specific to man and a condition that we are certain to obtain in the monkey), subjects will have to learn by trial and error during successive trials, the conditional associations between three abstract stimuli and three Manual responses (3 MRI-compatible mouse buttons).
Other: Second fMRI session — In this session (involving a condition specific to man and a condition that we are almost certain to obtain in monkeys), subjects will have to learn by trial and error during successive trials, the conditional associations between three abstract stimuli and Three orofacial responses (3 movements of the mouth).
Other: Third session of fMRI — In this session (involving a human-specific condition and a condition we hope to achieve in the monkey), subjects will have to learn by trial-error in successive trials, conditional associations between three abstract stimuli and three verbal or Vocals.

SUMMARY:
The cognitive control of speech is central to human social communication. Two frontal brain regions seem to have a critical role: 1) Broca's area (BA) and 2) the mid-cingulate cortex (MCC). Current rehabilitation strategy is clearly based on therapies promoting language performance. However, there is few evidence that rehabilitation strategies based on nonlinguistic aspects of brain function may enhance recovery. Such strategies may benefit from knowledge about the primary -nonlinguistic- function of the BA-MCC network. The aim of LANGUAGE is to identify this primary function. One hypothesis is that, in non-speaking primates, this network is involved in cognitive control of voluntary vocal/orofacial production. Specifically, whereas BA may be responsible for the high-level selection of orofacial and vocal responses during learning, the face motor representation within the MCC may be responsible for performance monitoring, a process inherently required in learning. LANGUAGE aims to test this hypothesis by determining in human the anatomo-functional organization of the BA-MCC network thanks to functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* being able to provide a written consent form
* having a social insurance
* have a normal vision (with or without corrections)
* Right-handed

Exclusion Criteria:

* Subjects with MRI contraindications (e.g. pacemaker, claustrophobia, metal in the body, etc…).
* Subjects must be willing to be advise in case of discovery of brain abnormality.
* History of known neurological or psychiatric illness
* Pregnant or nursing women
* Persons under guardianship, curators or any other administrative or judicial measure of deprivation of rights

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Behavioral data: performance in the task | 3 years
  Performance in the task will be assessed. If performance in the task is <80%, subjects will be excluded in the final analysis
fMRI data | 3 years
  BOLD signal will be analyzed in relation to the events of the task. Images must be not too much distorted to allow data analysis. As such, if a subject moved too much (translation>10mm; rotation>5°) the corresponding data will be excluded from the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Domenech, MD, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Hôpital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loh KK, Procyk E, Neveu R, Lamberton F, Hopkins WD, Petrides M, Amiez C. Cognitive control of orofacial motor and vocal responses in the ventrolateral and dorsomedial human frontal cortex. Proc Natl Acad Sci U S A. 2020 Mar 3;117(9):4994-5005. doi: 10.1073/pnas.1916459117. Epub 2020 Feb 14. PMID 32060124
- [Background] Loh KK, Hadj-Bouziane F, Petrides M, Procyk E, Amiez C. Rostro-Caudal Organization of Connectivity between Cingulate Motor Areas and Lateral Frontal Regions. Front Neurosci. 2018 Jan 11;11:753. doi: 10.3389/fnins.2017.00753. eCollection 2017. PMID 29375293
- [Background] Hillis AE. Magnetic resonance perfusion imaging in the study of language. Brain Lang. 2007 Aug;102(2):165-75. doi: 10.1016/j.bandl.2006.04.016. Epub 2006 Jun 6. PMID 16757020